CLINICAL TRIAL: NCT04566601
Title: A Phase II Randomized, Double-blinded, Placebo-controlled Parallel Group Trial to Examine the Efficacy and Safety of 4 Oral Doses of BI 1358894 Once Daily Over 12 Week Treatment Period in Patients With Borderline Personality Disorder
Brief Title: A Study to Test Different Doses of BI 1358894 and Find Out Whether They Reduce Symptoms in People With Borderline Personality Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1402-0012; 2020-000078-12 (EudraCT Number)
Record Dates: First submitted 2020-09-23; First posted 2020-09-28 (Actual); Results first posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Borderline Personality Disorder
MeSH Terms: conditions — Borderline Personality Disorder | interventions — TRPC inhibitor BI 1358894

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- BI 1358894 5mg (Experimental)
  Interventions: Drug: BI 1358894
- BI 1358894 25mg (Experimental)
  Interventions: Drug: BI 1358894
- BI 1358894 75mg (Experimental)
  Interventions: Drug: BI 1358894
- BI 1358894 125mg (Experimental)
  Interventions: Drug: BI 1358894
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 1358894 — Film-coated tablet
  Arms: BI 1358894 125mg; BI 1358894 25mg; BI 1358894 5mg; BI 1358894 75mg
Drug: Placebo — Film-coated tablet
  Arms: Placebo

SUMMARY:
This study is open to adults with borderline personality disorder. The purpose of this study is to find out whether a medicine called BI 1358894 helps to reduce symptoms in people with borderline personality disorder. Four different doses of BI 1358894 are tested in the study.

Participants are put into 5 groups by chance. Participants in 4 of the 5 groups take different doses of BI 1358894. Participants in the fifth group take placebo. Participants take BI 1358894 and placebo as tablets once a day. Placebo tablets look like BI 1358894 tablets but do not contain any medicine.

Participants are in the study for about 5 months. During this time, they visit the study site about 12 times and get about 6 phone calls. At the visits, doctors ask participants about their symptoms. The results between the BI 1358894 groups and the placebo group are then compared. The doctors also regularly check the general health of the participants.

ELIGIBILITY:
Inclusion Criteria:

* Patients meeting diagnostic criteria of borderline personality disorder (BoPD) per Diagnostic and Statistical Manual of Mental Disorders(DSM-5) at screening visit, confirmed by Structured Interview for DSM-5 Personality Disorder (SCID-5-PD).
* Zanarini rating scale for Borderline personality disorder (ZAN-BPD) of ≥ 9 at screening (Visit 1) and randomization (Visit 2), with question #2 Affective Instability score of ≥2.
* Male or female patients, 18-65 years of age at the time of consent
* Women of childbearing potential (WOCBP) able and willing to use two methods of contraception, as confirmed by the investigator, which include one highly effective method of birth control per ICH M3 (R2) that results in a low failure rate of less than 1%, plus one barrier method.

  --A woman is considered of childbearing potential (WOCBP), i.e. fertile, following menarche and until becoming postmenopausal unless permanently sterile. Permanent sterilization methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy. Tubal occlusion/ ligation is NOT a method of permanent sterilization. A postmenopausal state is defined as no menses for 12 months without an alternative medical cause.
* Signed and dated written informed consent in accordance with International Council on Harmonization (ICH) - Good Clinical Practice (GCP) and local legislation prior to admission to the trial.
* further inclusion criteria apply.

Exclusion Criteria:

* Current diagnosis of paranoid, schizoid, schizotypal and antisocial personality disorders, as confirmed by SCID-5-PD at screening visit.
* Lifetime diagnosis for schizophrenia, schizoaffective disorder, schizophreniform disorder, bipolar I disorder, or delusional disorder as confirmed by the SCID-5 at the screening visit.
* Any other mental disorder that is the primary focus of treatment in the last 6 months prior to randomization, as per the clinical judgement of the investigator.
* Inpatient stay or hospitalization due to worsening of BoPD within 3 months prior to randomization.
* Initiation or change in any type or frequency of psychotherapy for BoPD within the last 3 months prior to screening.
* Any ongoing use of psychotropic medications within 7 days prior to randomization or during the course of study.
* Any suicidal behavior in the past 1 year.
* Any suicidal ideation of type 4 or 5 in the Columbia Suicidal Severity Rating Scale (C-SSRS) in the past 3 months.
* further exclusion criteria apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Actual)
Dates: Start 2020-11-13 (Actual); Primary Completion 2022-12-09 (Actual); Study Completion 2023-01-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (67):
- United States (16):
  - Advanced Research Center, Inc., Anaheim, California
  - Viking Clinical Research, Ltd., Temecula, California
  - Pacific Clinical Research Management Group LLC, Upland, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Gulf Coast Clinical Research Center, Fort Myers, Florida
  - Sarkis Clinical Trials, Gainesville, Florida
  - San Marcus Research Clinic, Inc., Miami, Florida
  - Institute for Advanced Medical Research, Alpharetta, Georgia
  - McLean Hospital, Belmont, Massachusetts
  - Precise Research Centers, Flowood, Mississippi
  - Center For Emotional Fitness, Cherry Hill, New Jersey
  - University at Buffalo, The State University of New York, Buffalo, New York
  - Neurobehavioral Research, Inc., Cedarhurst, New York
  - Central States Research, LLC, Tulsa, Oklahoma
  - Grayline Research Center, Wichita Falls, Texas
  - Core Clinical Research, Everett, Washington
- Argentina (9):
  - Fundación para el Estudio y Tratamiento de las Enfermedades Mentales (FETEM), CABA
  - Fundación FunDaMos para la asistencia e investigación en psiquiatría, CABA
  - CEN (Centro Especializado Neurociencias), Córdoba
  - Instituto Modelo de Neurología Lennox, Córdoba
  - Instituto Médico DAMIC S.R.L., Córdoba
  - Clinica Privada de Salud Mental Santa Teresa de Avila, La Plata
  - Instituto de Neurociencias San Agustín, La Plata
  - Instituto Médico de la Fundación Estudios Clínicos, Rosario
  - Centro de Investigacion y Asistencia en Psiquiatria (CIAP), Rosario
- Australia (2):
  - Peninsula Therapeutic and Research Group, Frankston, Victoria
  - Monash Alfred Psychiatry Research Centre, Melbourne, Victoria
- Universitair Psychiatrisch Centrum Duffel (UPC Duffel), Duffel, Belgium
- Bulgaria (3):
  - "Filipopolis" - Ambulatory for Group Practice for Specialized Care in Psychiatry, Plovdiv
  - University Multiprofile Hospital for Active Treatement "Alexandrovska" EAD, Sofia
  - Medical Center Intermedica Ltd., Sofia
- Czechia (3):
  - MPMeditrine s.r.o., Ostrava-Poruba
  - Clintrial s.r.o., Prague
  - INEP medical s.r.o., Prague
- Denmark (2):
  - Aalborg Universitetsshospital, Aalborg
  - Region Zealand, Psychiatric Research Unit, Slagelse
- France (2):
  - HOP Pierre Wertheimer, Bron
  - HOP la Colombière, Montpellier
- Germany (7):
  - Universitätsklinikum Aachen, AöR, Aachen
  - Charité - Universitätsmedizin Berlin, Berlin
  - Universitätsklinikum Bonn AöR, Bonn
  - Universitätsklinikum Gießen und Marburg GmbH, Giessen
  - Zentralinstitut für seelische Gesundheit, Mannheim
  - Klinikum der Universität München - Campus Innenstadt, München
  - Universitätsklinikum Tübingen, Tübingen
- IRCCS San Giovanni Di Dio Fatebenefratelli, Brescia, Italy
- Japan (7):
  - Kokoro no Clinic Hirao, Fukuoka, Fukuoka
  - Hirota Clinic, Fukuoka, Kurume
  - Kishiro Mental Clinic, Kanagawa, Kawasaki
  - Hiyoshi Hospital, Kanagawa, Yokohama
  - Nara Medical University Hospital, Nara, Kashihara
  - i Kokoro Clinic Nihonbashi, Tokyo, Chuo-ku
  - Ichigaya Himorogi Clinic, Tokyo, Shinjuku-ku
- Mexico (6):
  - GabiPros S.C., Mexico City
  - Medical Care & Research SA de CV, Mérida
  - Hospital Universitario Dr Jose Eleuterio Gonzalez, Monterrey
  - CIT-Neuropsique S.C, Monterrey
  - Centro de Estudios Clinicos de Queretaro S.C, Querétaro
  - BIND Investigaciones S.C., San Luis Potosí City
- Poland (2):
  - Podlassian Center of Psychogeriatry, Bialystok, Bialystok
  - PI HOUSE Sp. z o.o., Gdansk, Gdansk
- Spain (3):
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Virgen del Rocío, Seville
  - CS Casa del Barco, Valladolid
- Sweden (3):
  - Psykiatri Södra Stockholm, Enskede
  - Sahlgrenska Universitetssjukhuset, Östra, Gothenburg
  - Akademiska sjukhuset, Uppsala

IPD SHARING:
Plan to Share IPD: Yes
After the study is completed and the primary manuscript is accepted for publishing, researchers can use this following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement". Also, Researchers can use the following link https://www.mystudywindow.com/msw/datasharing to find information in order to request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website. The data shared are the raw clinical study data sets.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'.For study data - 1. after the submission and approval of the research proposal (checks will be performed by both the independent review panel and the sponsor, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a 'Data Sharing Agreement'.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- [Derived] Dwyer JB, Schmahl C, Makinodan M, Fineberg SK, Sommer S, Wruck J, Jelaska A, Adeniji A, Goodman M. Efficacy and Safety of BI 1358894 in Patients With Borderline Personality Disorder: Results of a Phase 2 Randomized, Placebo-Controlled, Parallel Group Dose-Ranging Trial. J Clin Psychiatry. 2025 Jan 13;86(1):24m15523. doi: 10.4088/JCP.24m15523. PMID 39832346
- [Derived] Stoffers-Winterling JM, Storebo OJ, Pereira Ribeiro J, Kongerslev MT, Vollm BA, Mattivi JT, Faltinsen E, Todorovac A, Jorgensen MS, Callesen HE, Sales CP, Schaug JP, Simonsen E, Lieb K. Pharmacological interventions for people with borderline personality disorder. Cochrane Database Syst Rev. 2022 Nov 14;11(11):CD012956. doi: 10.1002/14651858.CD012956.pub2. PMID 36375174
- See also: Related Info — https://www.mystudywindow.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a Phase II, 12-week multicenter, multinational, randomised, double-blind, placebo-controlled, parallel-group trial in patients with borderline personality disorder (BPD). Eligible patients with BPD were randomised to receive either BI 1358894 or placebo in a 2.5:1:1:1:2 ratio (placebo or BI 1358894 5 milligram (mg), 25 mg, 75 mg, or 125 mg), for 12 weeks.
  This trial included a screening period, a 12-week randomised treatment period, and a 4-week follow-up period.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- Placebo: Patients were also administered for 12 weeks once daily, orally one film-coated tablet of placebo matching BI 1358894 5 milligram (mg), one film-coated tablet of placebo matching BI 1358894 25 mg and two film-coated tablets of placebo matching BI 1358894 50 mg.
- BI 1358894 5mg: Patients were administered for 12 weeks once daily, orally one film-coated tablet of 5 milligram (mg) of BI 1358894. In order to maintain blinding in regard to each treatment group since BI 1358894 tablets (5 mg, 25 mg, 50 mg) are different sizes, patients were also administered for 12 weeks once daily, orally one film-coated tablet of placebo matching BI 1358894 25 mg and two film-coated tablets of placebo matching BI 1358894 50 mg.
- BI 1358894 25mg: Patients were administered for 12 weeks once daily, orally one film-coated tablet of 25 milligram (mg) of BI 1358894. In order to maintain blinding in regard to each treatment group since BI 1358894 tablets (5 mg, 25 mg, 50 mg) are different sizes, patients were also administered for 12 weeks once daily, orally one film-coated tablet of placebo matching BI 1358894 5 mg and two film-coated tablets of placebo matching BI 1358894 50 mg.
- BI 1358894 75mg: Patients were administered for 12 weeks once daily, orally one film-coated tablet of 25 milligram (mg) of BI 1358894 and one film-coated tablet of 50 milligram (mg) of BI 1358894 (total BI 1358894 dose=75 mg). In order to maintain blinding in regard to each treatment group since BI 1358894 tablets (5 mg, 25 mg, 50 mg) are different sizes, patients were also administered for 12 weeks once daily, orally one film-coated tablet of placebo matching BI 1358894 5 mg and one film-coated tablet of placebo matching BI 1358894 50 mg.
- BI 1358894 125mg: Patients were administered for 12 weeks once daily, orally one film-coated tablet of 25 milligram (mg) of BI 1358894 and two film-coated tablets of 50 milligram (mg) of BI 1358894 (total BI 1358894 dose=125 mg). In order to maintain blinding in regard to each treatment group since BI 1358894 tablets (5 mg, 25 mg, 50 mg) are different sizes, patients were also administered for 12 weeks once daily, orally one film-coated tablet of placebo matching BI 1358894 5 mg.
Period: Overall Study
Arm/Group | Placebo | BI 1358894 5mg | BI 1358894 25mg | BI 1358894 75mg | BI 1358894 125mg
Started | 128 | 52 | 53 | 53 | 104
Completed (Completed planned trial treatment of 12 weeks.) | 95 | 40 | 35 | 40 | 77
Not Completed | 33 | 12 | 18 | 13 | 27
Not completed — Other than listed | 13 | 4 | 2 | 1 | 4
Not completed — Protocol deviation | 3 | 0 | 1 | 1 | 1
Not completed — Technical problems | 0 | 0 | 1 | 0 | 0
Not completed — No reason available | 3 | 2 | 7 | 1 | 5
Not completed — Burden of study procedures | 3 | 0 | 0 | 3 | 1
Not completed — Change of residence | 2 | 2 | 0 | 1 | 2
Not completed — Perceived lack of efficacy | 2 | 0 | 1 | 1 | 2
Not completed — Adverse Event | 7 | 4 | 6 | 5 | 12

BASELINE CHARACTERISTICS:
Population: Treated Set (TS) consisted of all patients who were randomised and that received at least one administration of trial medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | BI 1358894 5mg | BI 1358894 25mg | BI 1358894 75mg | BI 1358894 125mg | Total
Number analyzed (Participants) | 128 | 52 | 53 | 53 | 104 | 390
Age, Continuous [Mean (Standard Deviation); unit: Years] | 30.4 (9.9) | 29.2 (9.6) | 31.0 (11.1) | 30.6 (9.7) | 29.9 (11.2) | 30.2 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 107 | 50 | 48 | 48 | 83 | 336
  Male | 21 | 2 | 5 | 5 | 21 | 54
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 50 | 17 | 25 | 20 | 34 | 146
  Not Hispanic or Latino | 78 | 35 | 28 | 33 | 70 | 244
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 2 | 1 | 1 | 6 | 15
  Asian | 2 | 3 | 2 | 4 | 7 | 18
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 0 | 1
  Black or African American | 8 | 3 | 3 | 1 | 4 | 19
  White | 112 | 44 | 46 | 46 | 85 | 333
  More than one race | 0 | 0 | 1 | 1 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
ZAN-BPD total score at Baseline [Mean (Standard Deviation); unit: score on a scale] — The ZANarini rating scale for Borderline Personality Disorder (ZAN-BPD) reflects the nine DSM-5 (Diagnostic and Statistical Manual of Mental Disorders) criteria and the scale has 4 domain scores that reflect core areas of BPD (i.e., affective, cognitive, impulsive and interpersonal symptoms). The ZAN-BPD scale includes a 5-point rating scale (i.e., 0 = no symptoms to 4 = severe symptoms) for each criterion. The total ZAN-BPD score is the sum of the 4 domain scores and ranges from 0 to 36 where higher scores mean severe symptoms.
  score on a scale | 16.6 (5.0) | 15.7 (5.4) | 15.8 (4.8) | 16.1 (4.6) | 16.4 (5.2) | 16.3 (5.0)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in ZANarini Rating Scale for Borderline Personality Disorder (ZAN-BPD) Total Score at Week 10
Description: The ZAN-BPD scale reflects the nine DSM-5 criteria and the scale has 4 domain scores that reflect core areas of BPD (i.e., affective, cognitive, impulsive and interpersonal symptoms). The ZAN-BPD scale includes a 5-point rating scale (i.e., 0 = no symptoms to 4 = severe symptoms) for each criterion. The total ZAN-BPD score is the sum of the 4 domain scores and ranges from 0 to 36 where higher scores mean severe symptoms.
  Least Squares (LS) mean and standard error were estimated by restricted maximum likelihood-based mixed effects model repeated measures (REML-based MMRM) including the fixed categorical covariates of treatment, visit (baseline and Week 1, 2, 4, 6, 8 and 10) and the baseline ZAN-BPD total score strata indicator (<=18 vs. >=19), the continuous fixed covariate of baseline ZAN-BPD total score, and treatment-by-visit interaction, as well as baseline-by-visit interaction. LS mean (standard error) for Week 10 are reported.
Time Frame: The change from baseline at Week 10 in the total ZAN-BPD score was calculated using the MMRM model which is a longitudinal analyses and it incorporates ZAN-BPD measurements from baseline, Weeks 1, 2, 4, 6, 8 and Week 10.
Population: Full analysis set (FAS) consisted of all patients in TS who had a baseline and at least one evaluable post-baseline measurement for the primary endpoint. Since the MMRM included the measurements from baseline, Week 1, Week 2, Week 4, Week 6, Week 8 and Week 10, number of participants analyzed for the primary endpoint for each arm are the participants who had a ZAN-BPD score value at baseline and one ZAN-BPD score value at one of the post-baseline timepoints up to Week 10.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | BI 1358894 5mg | BI 1358894 25mg | BI 1358894 75mg | BI 1358894 125mg
Number analyzed (Participants) | 124 | 52 | 52 | 52 | 102
units on a scale | -8.7 (0.5) | -8.0 (0.9) | -9.2 (0.9) | -8.9 (0.8) | -9.0 (0.6)
Statistical Analysis 1: Comparison: Placebo vs BI 1358894 5mg; Least Squares (LS) mean difference and 95 % confidence interval were estimated by REML-based MMRM including the fixed categorical covariates of treatment, visit (baseline and Week 1, 2, 4, 6, 8, 10) and the baseline ZAN-BPD total score strata indicator (<=18 vs. >=19), the continuous fixed covariate of baseline ZAN-BPD total score, and treatment-by-visit interaction, as well as baseline-by-visit interaction. LS means differences (95 % confidence intervals) for Week 10 are reported; Test type: Other — No formal hypotheses were tested; p = 0.4994, Mixed effects model repeated measures — P-value is considered nominal; Mean Difference (Net) = 0.7, 95% CI 2-sided [-1.31 to 2.69] — Least Squares Mean of "BI 1358894 5mg" - Least Squares Mean of "Placebo"
Statistical Analysis 2: Comparison: Placebo vs BI 1358894 25mg; [analysis description as in outcome 1, analysis 1]; Test type: Other — No formal hypotheses were tested; p = 0.6014, Mixed effects model repeated measures — P-value is considered nominal; Mean Difference (Net) = -0.6, 95% CI 2-sided [-2.60 to 1.51] — Least Squares Mean of "BI 1358894 25mg" - Least Squares Mean of "Placebo"
Statistical Analysis 3: Comparison: Placebo vs BI 1358894 75mg; [analysis description as in outcome 1, analysis 1]; Test type: Other — No formal hypotheses were tested; p = 0.8166, Mixed effects model repeated measures — P-value is considered nominal; Mean Difference (Net) = -0.2, 95% CI 2-sided [-2.17 to 1.72] — Least Squares Mean of "BI 1358894 75mg" - Least Squares Mean of "Placebo"
Statistical Analysis 4: Comparison: Placebo vs BI 1358894 125mg; [analysis description as in outcome 1, analysis 1]; Test type: Other — No formal hypotheses were tested; p = 0.6588, Mixed effects model repeated measures — P-value is considered nominal; Mean Difference (Net) = -0.4, 95% CI 2-sided [-1.96 to 1.24] — Least Squares Mean of "BI 1358894 125mg" - Least Squares Mean of "Placebo"
Statistical Analysis 5: Comparison: Placebo vs BI 1358894 5mg vs BI 1358894 25mg vs BI 1358894 75mg vs BI 1358894 125mg; A flat vs. non-flat dose-response relationship across the 4 doses of BI 1358894 and placebo was tested using the Multiple Comparison Procedure - Modelling (MCP-Mod) approach which evaluated simultaneously 5 different plausible dose-response patterns (linear, exponential, Emax 1, Emax 2 and Sigmoid Emax) while protecting the overall probability of type I error (one-sided alpha of 0.100); Test type: Other — MMRM estimates were used as input for the MCP-Mod. MMRM included the fixed categorical covariates of treatment, visit (baseline and Week 1, 2, 4, 6, 8, 10) and the baseline ZAN-BPD total score strata indicator (<=18 vs. >=19), the continuous fixed covariate of baseline ZAN-BPD total score, and treatment-by-visit interaction, as well as baseline-by-visit interaction; p = 0.3914, MCP-Mod sigmoid Emax model fit; Model assumption: 50% of the maximum effect is achieved at 25 mg, and 90% of the maximum effect is achieved at 75 mg
Statistical Analysis 6: Comparison: Placebo vs BI 1358894 5mg vs BI 1358894 25mg vs BI 1358894 75mg vs BI 1358894 125mg; [analysis description as in outcome 1, analysis 5]; Test type: Other — MMRM estimates were used as input for the MCP-Mod. MMRM included the fixed categorical covariates of treatment, visit (baseline and Week 1, 2, 4, 6, 8, 10 and 12) and the baseline ZAN-BPD total score strata indicator (<=18 vs. >=19), the continuous fixed covariate of baseline ZAN-BPD total score, and treatment-by-visit interaction, as well as baseline-by-visit interaction; p = 0.4104, MCP-Mod Emax1 model fit; Model assumption: 50% of the maximum effect is achieved at 25 mg
Statistical Analysis 7: Comparison: Placebo vs BI 1358894 5mg vs BI 1358894 25mg vs BI 1358894 75mg vs BI 1358894 125mg; [analysis description as in outcome 1, analysis 5]; Test type: Other — [test comment as in outcome 1, analysis 5]; p = 0.4560, MCP-Mod linear model fit; Model assumption: No parameter assumptions required
Statistical Analysis 8: Comparison: Placebo vs BI 1358894 5mg vs BI 1358894 25mg vs BI 1358894 75mg vs BI 1358894 125mg; [analysis description as in outcome 1, analysis 5]; Test type: Other — [test comment as in outcome 1, analysis 5]; p = 0.4908, MCP-Mod exponential model fit; Model assumption: 5% of the maximum effect is achieved at 25 mg
Statistical Analysis 9: Comparison: Placebo vs BI 1358894 5mg vs BI 1358894 25mg vs BI 1358894 75mg vs BI 1358894 125mg; [analysis description as in outcome 1, analysis 5]; Test type: Other — [test comment as in outcome 1, analysis 5]; p = 0.4974, MCP-Mod Emax2 model fit; Model assumption: 70% of the maximum effect is achieved at 5 mg

2. Secondary Outcome: ZANarini Rating Scale for Borderline Personality Disorder (ZAN-BPD) Response: Defined as ≥30% ZAN-BPD Reduction From Baseline at Week 10
Description: Number of participants with ZAN-BPD response is reported. ZAN-BPD response was defined as ≥30% ZAN-BPD reduction from baseline at Week 10.
  The ZAN-BPD scale reflects the nine DSM-5 criteria, and the scale has 4 domain scores that reflect core areas of BPD (i.e., affective, cognitive, impulsive and interpersonal symptoms). The ZAN-BPD scale includes a 5-point rating scale (i.e., 0 = no symptoms to 4 = severe symptoms) for each criterion. The total ZAN-BPD score is the sum of the 4 domain scores and ranges from 0 to 36 where higher scores mean severe symptoms.
Time Frame: Baseline and at Week 10.
Population: Full analysis set (FAS) consisted of all patients in TS who had a baseline and at least one evaluable post-baseline measurement for the primary endpoint.
  Only participants with ZAN-BPD total score at baseline and at Week 10 are reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | BI 1358894 5mg | BI 1358894 25mg | BI 1358894 75mg | BI 1358894 125mg
Number analyzed (Participants) | 92 | 37 | 33 | 41 | 74
Participants | 68 | 22 | 28 | 34 | 59
Statistical Analysis 1: Comparison: Placebo vs BI 1358894 5mg; The odds ratio (OR) and associated confidence intervals between the active treatment arm versus placebo were calculated through a logistic regression model that was adjusted for fixed factors of treatment, baseline ZAN-BPD strata indicator (≤18 vs. ≥19), and the continuous covariate of baseline ZAN-BPD total score; Test type: Other; Odds Ratio (OR) = 0.486, 95% CI 2-sided [0.207 to 1.140] — Odds Ratio of BI 1358894 5mg vs. Placebo
Statistical Analysis 2: Comparison: Placebo vs BI 1358894 25mg; [analysis description as in outcome 2, analysis 1]; Test type: Other; Odds Ratio (OR) = 2.294, 95% CI 2-sided [0.829 to 7.480] — Odds Ratio of BI 1358894 25mg vs. Placebo
Statistical Analysis 3: Comparison: Placebo vs BI 1358894 75mg; [analysis description as in outcome 2, analysis 1]; Test type: Other; Odds Ratio (OR) = 1.753, 95% CI 2-sided [0.698 to 4.861] — Odds Ratio of BI 1358894 75mg vs. Placebo
Statistical Analysis 4: Comparison: Placebo vs BI 1358894 125mg; [analysis description as in outcome 2, analysis 1]; Test type: Other; Odds Ratio (OR) = 1.352, 95% CI 2-sided [0.642 to 2.913] — Odds Ratio of BI 1358894 125mg vs. Placebo

3. Secondary Outcome: Change From Baseline in Difficulties in Emotion Regulation Scale (DERS-16) Total Score at Week 10
Description: The DERS is a self-report measure of emotion regulation difficulties. It consists of 16 items that assess non-acceptance of negative emotions, inability to engage in goal-directed behaviors when distressed, difficulties controlling impulsive behaviors when distressed, limited access to emotion regulation strategies perceived as effective, and lack of emotional clarity. Each item is scored from 1 (almost never (0-10%)) to 5 (almost always (91-100%)). Total DERS-16 can range from 16 to 80, with higher scores reflecting greater levels of emotion dysregulation.
  Least Squares (LS) mean and standard error were estimated by REML-based MMRM including the fixed categorical covariates of treatment, visit (baseline and Week 1, 2, 4, 6, 8 and 10) and the continuous fixed covariate of baseline DERS-16 total score, and treatment-by-visit interaction, as well as baseline-by-visit interaction. Patient was considered as random. LS mean (standard error) for Week 10 are reported.
Time Frame: Change from baseline in DERS-16 total score at Week 10 was calculated using the MMRM model which is a longitudinal analyses and it incorporates DERS-16 measurements from baseline, Weeks 1, 2, 4, 6, 8 and Week 10.
Population: Full analysis set (FAS) consisted of all patients in TS who had a baseline and at least one evaluable post-baseline measurement for the primary endpoint. Since the MMRM included the measurements from baseline, Week 1, Week 2, Week 4, Week 6, Week 8 and Week 10, number of participants analyzed for the primary endpoint for each arm are the participants who had a DERS-16 total score value at baseline and a DERS-16 total score value at one of the post-baseline timepoints up to Week 10.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | BI 1358894 5mg | BI 1358894 25mg | BI 1358894 75mg | BI 1358894 125mg
Number analyzed (Participants) | 124 | 52 | 52 | 52 | 102
units on a scale | -9.77 (1.4) | -9.87 (2.1) | -9.76 (2.2) | -10.56 (2.1) | -8.60 (1.5)
Statistical Analysis 1: Comparison: Placebo vs BI 1358894 5mg; Least Squares (LS) mean difference and 95% confidence interval were estimated by REML-based MMRM including the fixed categorical covariates of treatment, visit (baseline and Week 1, 2, 4, 6, 8, 10) and the continuous fixed covariate of baseline DERS-16 total score, and treatment-by-visit interaction, as well as baseline-by-visit interaction. Patient was considered as random. Unstructured covariance matrix was used; Test type: Other — No formal hypotheses were tested; p = 0.9675, Mixed effects model repeated measures — P-value is considered nominal; Mean Difference (Net) = -0.10, 95% CI 2-sided [-5.11 to 4.90] — Least Squares Mean of "BI 1358894 5mg" - Least Squares Mean of "Placebo"
Statistical Analysis 2: Comparison: Placebo vs BI 1358894 25mg; [analysis description as in outcome 3, analysis 1]; Test type: Other — No formal hypotheses were tested; p = 0.9969, Mixed effects model repeated measures — P-value is considered nominal; Mean Difference (Net) = 0.01, 95% CI 2-sided [-5.08 to 5.10] — Least Squares Mean of "BI 1358894 25mg" - Least Squares Mean of "Placebo"
Statistical Analysis 3: Comparison: Placebo vs BI 1358894 75mg; [analysis description as in outcome 3, analysis 1]; Test type: Other — No formal hypotheses were tested; p = 0.7542, Mixed effects model repeated measures — P-value is considered nominal; Mean Difference (Net) = -0.79, 95% CI 2-sided [-5.73 to 4.15] — Least Squares Mean of "BI 1358894 75mg" - Least Squares Mean of "Placebo"
Statistical Analysis 4: Comparison: Placebo vs BI 1358894 125mg; [analysis description as in outcome 3, analysis 1]; Test type: Other — No formal hypotheses were tested; p = 0.5683, Mixed effects model repeated measures — P-value is considered nominal; Mean Difference (Net) = 1.17, 95% CI 2-sided [-2.86 to 5.19] — Least Squares Mean of "BI 1358894 125mg" - Least Squares Mean of "Placebo"

4. Secondary Outcome: Change From Baseline in State-Trait Anxiety Inventory (STAI-S) Total Score at Week 10
Description: The STAI-S consists of 20 item state anxiety questions that evaluate how respondents feel "right now, at this moment". All items are rated on a weighted score of 1 to 4 scale (e.g. from 'Almost Never to 'Almost Always'); with higher scores indicating greater anxiety. STAI-S score ranges from 20 to 80 where higher scores indicate greater anxiety.
  Least Squares (LS) mean and standard error were estimated by restricted maximum likelihood-based mixed effects model repeated measures (REML-based MMRM) including the fixed categorical covariates of treatment, visit (baseline and Week 1, 2, 4, 6, 8, 10) and the continuous fixed covariate of baseline STAI-S total score, and treatment-by-visit interaction, as well as baseline-by-visit interaction. Patient was considered as random. LS mean (standard error) for Week 10 are reported.
Time Frame: Change from baseline in STAI-S total score at Week 10 was calculated using the MMRM model which is a longitudinal analyses and it incorporates STAI-S measurements from baseline, Weeks 1, 2, 4, 6, 8 and Week 10.
Population: Full analysis set (FAS) consisted of all patients in TS who had a baseline and at least one evaluable post-baseline measurement for the primary endpoint. Since the MMRM included the measurements from baseline, Week 1, Week 2, Week 4, Week 6, Week 8 and Week 10, number of participants analyzed for the primary endpoint for each arm are the participants who had a STAI-S total score value at baseline and a STAI-S total score value at one of the post-baseline timepoints up to Week 10.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | BI 1358894 5mg | BI 1358894 25mg | BI 1358894 75mg | BI 1358894 125mg
Number analyzed (Participants) | 124 | 52 | 52 | 52 | 102
units on a scale | -6.64 (1.2) | -8.71 (1.9) | -5.43 (2.0) | -7.00 (1.8) | -5.49 (1.3)
Statistical Analysis 1: Comparison: Placebo vs BI 1358894 5mg; Least Squares (LS) mean difference and 95% confidence interval were estimated by restricted maximum likelihood-based mixed effects model repeated measures (REML-based MMRM) including the fixed categorical covariates of treatment, visit (baseline and Week 1, 2, 4, 6, 8, 10) and the continuous fixed covariate of baseline STAI-S total score, and treatment-by-visit interaction, as well as baseline-by-visit interaction. Patient was considered as random. Unstructured covariance matrix was used; Test type: Other — No formal hypotheses were tested; p = 0.3568, Mixed effects model repeated measures — P-value is considered nominal; Mean Difference (Net) = -2.07, 95% CI 2-sided [-6.49 to 2.35] — Least Squares Mean of "BI 1358894 5mg" - Least Squares Mean of "Placebo"
Statistical Analysis 2: Comparison: Placebo vs BI 1358894 25mg; [analysis description as in outcome 4, analysis 1]; Test type: Other — No formal hypotheses were tested; p = 0.6009, Mixed effects model repeated measures — P-value is considered nominal; Mean Difference (Net) = 1.21, 95% CI 2-sided [-3.33 to 5.75] — Least Squares Mean of "BI 1358894 25mg" - Least Squares Mean of "Placebo"
Statistical Analysis 3: Comparison: Placebo vs BI 1358894 75mg; [analysis description as in outcome 4, analysis 1]; Test type: Other — No formal hypotheses were tested; p = 0.8705, Mixed effects model repeated measures — P-value is considered nominal; Mean Difference (Net) = -0.36, 95% CI 2-sided [-4.70 to 3.98] — Least Squares Mean of "BI 1358894 75mg" - Least Squares Mean of "Placebo"
Statistical Analysis 4: Comparison: Placebo vs BI 1358894 125mg; [analysis description as in outcome 4, analysis 1]; Test type: Other — No formal hypotheses were tested; p = 0.5262, Mixed effects model repeated measures — P-value is considered nominal; Mean Difference (Net) = 1.15, 95% CI 2-sided [-2.41 to 4.71] — Least Squares Mean of "BI 1358894 125mg" - Least Squares Mean of "Placebo"

5. Secondary Outcome: Change From Baseline in Patient Health Questionnaire (PHQ-9) Total Score at Week 10
Description: The PHQ-9 is a 9-item brief self-reported tool used for screening, diagnosing, monitoring and measuring the severity of depression. PHQ-9 has a maximum total score of 27. Depression Severity is assessed as: none (0-4), mild (5-9), moderate (10-14), moderately severe (15-19), or severe (20-27).
  Least Squares (LS) mean and standard error were estimated by restricted maximum likelihood-based mixed effects model repeated measures (REML-based MMRM) including the fixed categorical covariates of treatment, visit (baseline and Week 1, 2, 4, 6, 8, 10) and the continuous fixed covariate of baseline PHQ-9 total score, and treatment-by-visit interaction, as well as baseline-by-visit interaction. Patient was considered as random. LS mean (standard error) for Week 10 are reported.
Time Frame: Change from baseline in PHQ-9 total score at Week 10 was calculated using the MMRM model which is a longitudinal analyses and it incorporates PHQ-9 measurements from baseline, Weeks 1, 2, 4, 6, 8 and Week 10.
Population: Full analysis set (FAS) consisted of all patients in TS who had a baseline and at least one evaluable post-baseline measurement for the primary endpoint. Since the MMRM included the measurements from baseline, Week 1, Week 2, Week 4, Week 6, Week 8 and Week 10, number of participants analyzed for the primary endpoint for each arm are the participants who had a PHQ-9 total score value at baseline and a PHQ-9 total score value at one of the post-baseline timepoints up to Week 10.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | BI 1358894 5mg | BI 1358894 25mg | BI 1358894 75mg | BI 1358894 125mg
Number analyzed (Participants) | 124 | 52 | 52 | 52 | 102
units on a scale | -1.30 (0.6) | -3.13 (0.9) | -1.07 (0.9) | -1.57 (0.9) | -1.43 (0.6)
Statistical Analysis 1: Comparison: Placebo vs BI 1358894 5mg; Least Squares (LS) mean difference and 95% confidence interval were estimated by restricted maximum likelihood-based mixed effects model repeated measures (REML-based MMRM) including the fixed categorical covariates of treatment, visit (baseline and Week 1, 2, 4, 6, 8, 10) and the continuous fixed covariate of baseline PHQ-9 total score, and treatment-by-visit interaction, as well as baseline-by-visit interaction. Patient was considered as random. Unstructured covariance matrix was used; Test type: Other — No formal hypotheses were tested; p = 0.0782, Mixed effects model repeated measures — P-value is considered nominal; Mean Difference (Net) = -1.83, 95% CI 2-sided [-3.87 to 0.21] — Least Squares Mean of "BI 1358894 5mg" - Least Squares Mean of "Placebo"
Statistical Analysis 2: Comparison: Placebo vs BI 1358894 25mg; [analysis description as in outcome 5, analysis 1]; Test type: Other — No formal hypotheses were tested; p = 0.8266, Mixed effects model repeated measures — P-value is considered nominal; Mean Difference (Net) = 0.23, 95% CI 2-sided [-1.86 to 2.32] — Least Squares Mean of "BI 1358894 25mg" - Least Squares Mean of "Placebo"
Statistical Analysis 3: Comparison: Placebo vs BI 1358894 75mg; [analysis description as in outcome 5, analysis 1]; Test type: Other — No formal hypotheses were tested; p = 0.7910, Mixed effects model repeated measures — P-value is considered nominal; Mean Difference (Net) = -0.27, 95% CI 2-sided [-2.28 to 1.74] — Least Squares Mean of "BI 1358894 75mg" - Least Squares Mean of "Placebo"
Statistical Analysis 4: Comparison: Placebo vs BI 1358894 125mg; [analysis description as in outcome 5, analysis 1]; Test type: Other — No formal hypotheses were tested; p = 0.8743, Mixed effects model repeated measures — P-value is considered nominal; Mean Difference (Net) = -0.13, 95% CI 2-sided [-1.77 to 1.51] — Least Squares Mean of "BI 1358894 125mg" - Least Squares Mean of "Placebo"

6. Secondary Outcome: Change From Baseline in Clinical Global Impression Severity Scale (CGI-S) at Week 10
Description: The CGI-S rating scale measures the clinician's impression of the severity of illness exhibited by a participant. The CGI-S only question states "Considering your total clinical experience with this particular population, please choose the response below that best describes how mentally ill the patient was over the past week?", and is rated on the following seven-point scale: 1=normal, not at all ill; 2=borderline ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; 7=among the most extremely ill patients.
  Least Squares (LS) mean and standard error were estimated by REML-based MMRM including the fixed categorical covariates of treatment, visit (baseline and Week 1, 2, 4, 6, 8, 10) and the continuous fixed covariate of baseline CGI-S total score, and treatment-by-visit interaction, as well as baseline-by-visit interaction. Patient was considered as random. LS mean (standard error) for Week 10 are reported.
Time Frame: Change from baseline in CGI-S scale at Week 10 was calculated using the MMRM model which is a longitudinal analyses and it incorporates CGI-S measurements from baseline, Weeks 1, 2, 4, 6, 8 and Week 10.
Population: Full analysis set (FAS) consisted of all patients in TS who had a baseline and at least one evaluable post-baseline measurement for the primary endpoint. Since the MMRM included the measurements from baseline, Week 1, Week 2, Week 4, Week 6, Week 8 and Week 10, number of participants analyzed for the primary endpoint for each arm are the participants who had a CGI-S scale value at baseline and a CGI-S scale value at one of the post-baseline timepoints up to Week 10.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | BI 1358894 5mg | BI 1358894 25mg | BI 1358894 75mg | BI 1358894 125mg
Number analyzed (Participants) | 124 | 52 | 51 | 51 | 102
units on a scale | -1.23 (0.1) | -1.29 (0.2) | -1.47 (0.2) | -1.24 (0.2) | -1.42 (0.1)
Statistical Analysis 1: Comparison: Placebo vs BI 1358894 5mg; Least Squares (LS) mean difference and 95% confidence interval were estimated by restricted maximum likelihood-based mixed effects model repeated measures (REML-based MMRM) including the fixed categorical covariates of treatment, visit (baseline and Week 1, 2, 4, 6, 8, 10) and the continuous fixed covariate of baseline CGI-S total score, and treatment-by-visit interaction, as well as baseline-by-visit interaction. Patient was considered as random. Unstructured covariance matrix was used; Test type: Other — No formal hypotheses were tested; p = 0.8016, Mixed effects model repeated measures — P-value is considered nominal; Mean Difference (Net) = -0.05, 95% CI 2-sided [-0.47 to 0.37] — Least Squares Mean of "BI 1358894 5mg" - Least Squares Mean of "Placebo"
Statistical Analysis 2: Comparison: Placebo vs BI 1358894 25mg; [analysis description as in outcome 6, analysis 1]; Test type: Other — No formal hypotheses were tested; p = 0.2929, Mixed effects model repeated measures — P-value is considered nominal; Mean Difference (Net) = -0.23, 95% CI 2-sided [-0.67 to 0.20] — Least Squares Mean of "BI 1358894 25mg" - Least Squares Mean of "Placebo"
Statistical Analysis 3: Comparison: Placebo vs BI 1358894 75mg; [analysis description as in outcome 6, analysis 1]; Test type: Other — No formal hypotheses were tested; p = 0.9666, Mixed effects model repeated measures — P-value is considered nominal; Mean Difference (Net) = -0.01, 95% CI 2-sided [-0.42 to 0.40] — Least Squares Mean of "BI 1358894 75mg" - Least Squares Mean of "Placebo"
Statistical Analysis 4: Comparison: Placebo vs BI 1358894 125mg; [analysis description as in outcome 6, analysis 1]; Test type: Other — No formal hypotheses were tested; p = 0.2833, Mixed effects model repeated measures — P-value is considered nominal; Mean Difference (Net) = -0.18, 95% CI 2-sided [-0.52 to 0.15] — Least Squares Mean of "BI 1358894 125mg" - Least Squares Mean of "Placebo"

7. Secondary Outcome: Change From Baseline in Patient Global Impression Severity Scale (PGI-S) at Week 10
Description: The PGI-S measures the patient's impression of the severity of their illness. It is a single item 5-point scale that asks patients to rate the severity of their illness. The PGI-S question states "Please choose the response below that best describes the overall severity of your symptoms of Borderline Personality Disorder at this time. (Select one response)": 1=No symptoms; 2=Mild; 3=Moderate; 4=Severe; 5=Very severe.
  Least Squares (LS) mean and standard error were estimated by restricted maximum likelihood-based mixed effects model repeated measures (REML-based MMRM) including the fixed categorical covariates of treatment, visit (baseline and Week 1, 2, 4, 6, 8,10) and the continuous fixed covariate of baseline PGI-S total score, and treatment-by-visit interaction, as well as baseline-by-visit interaction. Patient was considered as random. LS means (standard error) for Week 10 are reported.
Time Frame: Change from baseline in PGI-S scale at Week 10 was calculated using the MMRM model which is a longitudinal analyses and it incorporates PGI-S measurements from baseline, Weeks 1, 2, 4, 6, 8 and Week 10.
Population: Full analysis set (FAS) consisted of all patients in TS who had a baseline and at least one evaluable post-baseline measurement for the primary endpoint. Since the MMRM included the measurements from baseline, Week 1, Week 2, Week 4, Week 6, Week 8 and Week 10, number of participants analyzed for the primary endpoint for each arm are the participants who had a PGI-S scale value at baseline and a PGI-S scale value at one of the post-baseline timepoints up to Week 10.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | BI 1358894 5mg | BI 1358894 25mg | BI 1358894 75mg | BI 1358894 125mg
Number analyzed (Participants) | 124 | 52 | 50 | 52 | 102
units on a scale | -0.61 (0.1) | -0.73 (0.1) | -0.73 (0.2) | -0.64 (0.1) | -0.69 (0.1)
Statistical Analysis 1: Comparison: Placebo vs BI 1358894 5mg; Least Squares (LS) mean difference and 95% confidence interval were estimated by restricted maximum likelihood-based mixed effects model repeated measures (REML-based MMRM) including the fixed categorical covariates of treatment, visit (baseline and Week 1, 2, 4, 6, 8, 10) and the continuous fixed covariate of baseline PGI-S total score, and treatment-by-visit interaction, as well as baseline-by-visit interaction. Patient was considered as random. Unstructured covariance matrix was used; Test type: Other — No formal hypotheses were tested; p = 0.4552, Mixed effects model repeated measures — P-value is considered nominal; Mean Difference (Net) = -0.13, 95% CI 2-sided [-0.45 to 0.20] — Least Squares Mean of "BI 1358894 5mg" - Least Squares Mean of "Placebo"
Statistical Analysis 2: Comparison: Placebo vs BI 1358894 25mg; [analysis description as in outcome 7, analysis 1]; Test type: Other — No formal hypotheses were tested; p = 0.4734, Mixed effects model repeated measures — P-value is considered nominal; Mean Difference (Net) = -0.13, 95% CI 2-sided [-0.47 to 0.22] — Least Squares Mean of "BI 1358894 25mg" - Least Squares Mean of "Placebo"
Statistical Analysis 3: Comparison: Placebo vs BI 1358894 75mg; [analysis description as in outcome 7, analysis 1]; Test type: Other — No formal hypotheses were tested; p = 0.8388, Mixed effects model repeated measures — P-value is considered nominal; Mean Difference (Net) = -0.03, 95% CI 2-sided [-0.36 to 0.29] — Least Squares Mean of "BI 1358894 75mg" - Least Squares Mean of "Placebo"
Statistical Analysis 4: Comparison: Placebo vs BI 1358894 125mg; [analysis description as in outcome 7, analysis 1]; Test type: Other — No formal hypotheses were tested; p = 0.5540, Mixed effects model repeated measures — P-value is considered nominal; Mean Difference (Net) = -0.08, 95% CI 2-sided [-0.35 to 0.19] — Least Squares Mean of "BI 1358894 125mg" - Least Squares Mean of "Placebo"

ADVERSE EVENTS:
Time Frame: From first dose of study drug administration until the last dose of study drug administration + 4 weeks of residual effect period, up to 17 weeks.
Description: Treated set (TS) consisted of all patients who were randomised and that received at least 1 administration of trial medication. Patients were analysed according to the actual received treatment.
Arm/Group | Placebo | BI 1358894 5mg | BI 1358894 25mg | BI 1358894 75mg | BI 1358894 125mg
All-Cause Mortality (participants affected / at risk) | 0/128 | 0/52 | 0/53 | 0/53 | 2/104
Serious Adverse Events (participants affected / at risk) | 11/128 | 4/52 | 3/53 | 4/53 | 16/104
Other Adverse Events (participants affected / at risk) | 75/128 | 32/52 | 40/53 | 34/53 | 61/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=128) | BI 1358894 5mg (N=52) | BI 1358894 25mg (N=53) | BI 1358894 75mg (N=53) | BI 1358894 125mg (N=104)
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Cannabinoid hyperemesis syndrome (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Death (General disorders) | 0 | 0 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 0 | 0 | 1
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Hepatitis A (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Wound abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Comminuted fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Forearm fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 1
Aggression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Drug abuse (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Panic attack (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Post-traumatic stress disorder (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Suicidal behaviour (Psychiatric disorders) | 0 | 1 | 0 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 8 | 3 | 1 | 1 | 6
Suicide attempt (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Calculus urinary (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=128) | BI 1358894 5mg (N=52) | BI 1358894 25mg (N=53) | BI 1358894 75mg (N=53) | BI 1358894 125mg (N=104)
Constipation (Gastrointestinal disorders) | 2 | 2 | 5 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 10 | 4 | 3 | 3 | 4
Dyspepsia (Gastrointestinal disorders) | 1 | 2 | 1 | 3 | 0
Nausea (Gastrointestinal disorders) | 17 | 5 | 5 | 2 | 7
Fatigue (General disorders) | 11 | 6 | 1 | 6 | 9
Pyrexia (General disorders) | 2 | 4 | 3 | 2 | 1
COVID-19 (Infections and infestations) | 16 | 3 | 1 | 6 | 7
Influenza (Infections and infestations) | 8 | 3 | 1 | 1 | 7
Nasopharyngitis (Infections and infestations) | 10 | 3 | 3 | 7 | 9
Pharyngitis (Infections and infestations) | 2 | 3 | 0 | 0 | 0
Weight increased (Investigations) | 0 | 1 | 1 | 3 | 5
Hyperinsulinaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 3 | 0
Increased appetite (Metabolism and nutrition disorders) | 4 | 1 | 1 | 1 | 8
Disturbance in attention (Nervous system disorders) | 5 | 3 | 2 | 4 | 0
Dizziness (Nervous system disorders) | 9 | 6 | 5 | 7 | 8
Headache (Nervous system disorders) | 32 | 18 | 23 | 15 | 33
Somnolence (Nervous system disorders) | 4 | 3 | 5 | 6 | 4
Anxiety (Psychiatric disorders) | 9 | 6 | 3 | 3 | 3
Initial insomnia (Psychiatric disorders) | 5 | 1 | 0 | 3 | 0
Insomnia (Psychiatric disorders) | 10 | 5 | 5 | 4 | 6
Intentional self-injury (Psychiatric disorders) | 7 | 2 | 1 | 2 | 3
Dysmenorrhoea (Reproductive system and breast disorders) | 3 | 0 | 1 | 5 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 0 | 1 | 2 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 9 | 3 | 0 | 2 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2022-09-23): https://cdn.clinicaltrials.gov/large-docs/01/NCT04566601/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-26): https://cdn.clinicaltrials.gov/large-docs/01/NCT04566601/SAP_001.pdf